CLINICAL TRIAL: NCT00787657
Title: Betaferon Prospective Study on Adherence, Coping and Nursing Support
Brief Title: Observational Study to Analyse the Impact of Nurse Support and Disease Related Factors on Long- Term Adherence to Betaferon Treatment
Acronym: BEACON
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 13852; 311941 (Other: company internal); BF0703 (Other: company internal)
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis (RRMS)
Keywords: Clinically Isolated Syndrome (CIS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm 1
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Patients after first clinical events suggestive of MS (according to SMPC) and patients with RRMS within the first two years of diagnosis

SUMMARY:
* The Study analyses the influence of selected factors on adherence to Betaferon treatment in patients with early multiple sclerosis (MS). The Investigator will document the relevant medical data regarding multiple sclerosis at every hospital visit, the patient will fill in two questionnaires at every visit: one about coping with the disease and the other about anxiety and depression.
* The Study particularly looks at the role of the support of the patient given by the multiple sclerosis nurses.The nurse will provide additional standardised information at start of treatment and will regularly phone the patient to ask standardised questions about the general condition with regard to the treatment, the disease and social support. At the end of the Study it will be assessed if the supportive measures and the standards in terms of adherence management in the hospital have some influence to increase long-term treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patients after first clinical event suggestive of multiple Sclerosis (MS) (according to SmPC) and patients with Relapsing / Remitting Multiple Sclerosis (RRMS) within the first two years of diagnosis.

Exclusion Criteria:

* Contra-indications as indicated in Betaferon summary of Products Characteristics (SmPC)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients after clinical events suggestive of MS according to SMPC) and patients with elapsing / Remitting Multiple Sclerosis (RRMS) within the first two years of diagnosis
Sampling Method: Probability Sample
Enrollment: 1723 (Actual)
Dates: Start 2008-06; Primary Completion 2013-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients adhering to treatment | 6, 12, 18 and 24 months

SECONDARY OUTCOMES:
Rate of early treatment termination | 6, 12, 18 and 24 months
Rate of study dropout | 6, 12, 18 and 24 months
Predictive value of BL parameters, WCQ, HADS, RODQ | 12 and 24 months
WCQ (Ways of Coping Questionnaire) | 6, 12, 18 and 24 months
HADS (Hospital Anxiety and Depression Scale) | 6, 12, 18 and 24 months
RODQ (Risk of Dropout Questionnaire) | Monthly over 6 months; every other month thereafter
EDSS (Expanded Disability Status Scale) | 6, 12, 18 and 24 months
Relapse rate | 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (36):
- Many Locations, Argentina
- Many Locations, Bahrain
- Many Locations, Belgium
- Many Locations, Bosnia and Herzegovina
- Many Locations, Canada
- Many Locations, China
- Many Locations, Colombia
- Many Locations, Czechia
- Many Locations, Egypt
- Many Locations, Estonia
- Many Locations, France
- Many Locations, Germany
- Many Locations, Iran
- Many Locations, Israel
- Many Locations, Italy
- Many Locations, Jordan
- Many Locations, Kuwait
- Many Locations, Lebanon
- Many Locations, Libya
- Many Locations, Mexico
- Many Locations, Netherlands
- Many Locations, New Zealand
- Many Locations, Norway
- Many Locations, Pakistan
- Many Locations, Portugal
- Many Locations, Saudi Arabia
- Many Locations, Singapore
- Many Locations, Slovakia
- Many Locations, Slovenia
- Many Locations, South Korea
- Many Locations, Sweden
- Many Locations, Syria
- Many Locations, Taiwan
- Many Locations, United Arab Emirates
- Many Locations, United Kingdom
- Many Locations, Venezuela

REFERENCES:
- [Derived] Patti F, Penaherrera JN, Zieger L, Wicklein EM. Clinical characteristics of middle-aged and older patients with MS treated with interferon beta-1b: post-hoc analysis of a 2-year, prospective, international, observational study. BMC Neurol. 2021 Aug 23;21(1):324. doi: 10.1186/s12883-021-02347-w. PMID 34425763